CLINICAL TRIAL: NCT05351229
Title: Intrathecal Morphine for Postoperative Analgesia in Video-Assisted and Robotic-Assisted Thoracic Surgery: A Randomized, Placebo-controlled, Double-blinded Clinical Trial
Brief Title: Intrathecal Morphine for Analgesia in Video-assisted and Robotic-assisted Thoracic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richa Dhawan, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB22-0561
Record Dates: First submitted 2022-04-13; First posted 2022-04-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Intervention Model Description: Intervention is intrathecal morphine in the intervention group. The drug is PF morphine
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo, Intrathecal saline
  Interventions: Other: Placebo
- Morphine (Active Comparator): Intrathecal morphine
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Morphine Sulfate — 5 mcg/kg intrathecal preservative free morphine sulfate
  Arms: Morphine
Other: Placebo — Sterile saline, placebo
  Other Names: Sterile Saline
  Arms: Placebo

SUMMARY:
VATS/RATS is widely used for diagnosis and treatment of intrathoracic conditions. Despite many benefits, postoperative pain continues to be intense after VATS/RATS. The optimal strategy for pain management has not been defined. In this randomized, placebo-controlled, double-blinded clinical investigation, investigators hypothesize that 5 mcg/kg intrathecal morphine will decrease postoperative analgesic consumption and reduce pain.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blinded clinical trial. Patients will be randomized into one of two groups. Group A (Placebo, control group) will receive intrathecal sterile normal saline and Group B (Morphine group) will receive 5mcg/kg preservative free intrathecal morphine.

American Pain Society Outcome Questionnaire (APS-POQ) will be administered to patients prior to discharge (see data sheet).

Patients will be followed up with a phone survey at 1 and 3 months after surgery to assess the presence, nature, and severity of chronic persistent surgical pain. The Brief Pain Inventory is a reliable and valid measures of the interference of pain with physical functioning and will be used. Additionally patients will be asked about use of pain medications

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* Undergoing elective video-assisted thoracoscopic or robotic assisted surgery for anatomical lung resection
* General anesthesia with anticipated intraoperative extubation.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) classification of 4 or 5
* Anticipated postoperative intubation
* Significant liver disease
* Preoperative use of intravenous inotropes and/or vasopressor support
* Preoperative mechanical ventilation
* Preoperative use of mechanical circulatory support device (intraaortic balloon pump, ventricular assist device, extracorporeal membrane oxygenation)
* Severe pulmonary disease (home oxygen requirement and/or current oral steroid use)
* Morphine allergy
* Opioid or alcohol abuse
* Chronic pain
* Renal failure
* Inability to comprehend English language
* Bleeding disorder
* Abnormal preoperative coagulation
* Infection
* Patient refusal
* Failed spinal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative morphine equivalent consumption | 24 hours after surgery
  Total MG of analgesic medications given converted to morphine

SECONDARY OUTCOMES:
Postoperative pain | Up to 48 hours postoperative
  Visual analog score between 0-10
Number of pain interventions | up to 48 hours postoperative
  Number of times patient given medication for pain
Postoperative opioid related side effects | up to 48 hours postoperative
  Nausea medication administration, airway events, urinary retention, pruritus medication given,
Self-reported patient satisfaction | prior to discharge from hospital, likely 1-3 days after surgery
  American Pain Society Outcome Questionnaire
pain qualities | 1 month and 3 months after surgery
  pain intensity, location, quality via Brief Pain Inventory
Self reported use of analgesic medications | 1 month and 3 months after surgery
  Questions asked via phone call at 1 month and 3 months.
self-reported limitation of daily activity at 1 and 3 months | 1 month and 3 months after surgery
  Questions asked via phone call at 1 month and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Not necessary to conduct study or data analysis